CLINICAL TRIAL: NCT04043221
Title: Effects of Long Term Treatment With Metformin on Clinical, Metabolic and Endocrine Parameters in Women With Polycystic Ovary Syndrome And Increased Metabolic Risk
Brief Title: Long Term Metformin in Women With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, Clinical professor, University Medical Centre Ljubljana
Other Study IDs: MET retro
Record Dates: First submitted 2019-07-09; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators analyzed collection data of 10 years for the efficacy of metformin on body mass, menstrual frequencies, metabolic and hormonal outcomes in women with polycystic ovary syndrome (PCOS) and BMI ≥ 25kg/m2.

Each patient's age and height were recorded at baseline. In addition each patient weight, waist circumference, menstrual regularity, fasting glucose, glucose after 120 minute oral glucose tolerance test, luteinizing hormone, follicle stimulating hormone , free and direct testosterone, androstenedione, sex hormone binding globulin, dehydroepiandrosterone sulfate were identified at baseline and at the every follow up visit where available.

ELIGIBILITY:
Inclusion Criteria:

* PCOS phenotype A
* BMI≥ 25kg/m2
* metformin 1000mg twice a day for at least one year

Exclusion Criteria:

* PCOS phenotype B, C, D
* BMI <25kg/m2
* had been treated with spironolactone or oral contraceptives alone or in combination with metformin
* had history of bariatric surgery
* became pregnant during the observation period
* had inability to tolerate metformin, leading to the cessation of drug therapy within first follow up year

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Collection data from endocrine outpatient clinic for 10 years of women with PCOS phenotype A, BMI≥ 25kg/m2, all receiving monotherapy with metformin 1000 mg twice a day.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
body weight | The measurement is assessed in kilograms at the beginning and after every year of taking metformin for 10 years.
  Primary outcome was change in body weight.
menstrual frequency | The measurement is assessed in number of bleeds per year at the beginning and after every year of taking metformin for 10 years.
  Primary outcome was change in menstrual frequency.
free testosterone | The measurement is assessed in nmol/L at the beginning and after every year of taking metformin for 10 years.
  Primary outcome was change in levels of free testosterone.
diabetes mellitus | The measurement of glucose in blood is assessed in mmol/L at the beginning and after every year of taking metformin for 10 years.
  Primary outcome was development of diabetes mellitus.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia